CLINICAL TRIAL: NCT05314010
Title: A Multicenter, Phase Ib/III Study to Evaluate the Safety and Efficacy of MIL62 in Patients With Neuromyelitis Optica Spectrum Disorder (NMOSD)
Brief Title: A Study of MIL62 in Patients With Neuromyelitis Optica Spectrum Disorder (NMOSD)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing Mabworks Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MIL62-CT303
Record Dates: First submitted 2022-03-29; First posted 2022-04-06 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2024-10

CONDITIONS: Neuromyelitis Optica Spectrum Disorder
MeSH Terms: conditions — Neuromyelitis Optica

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MIL62 (Experimental)
  Interventions: Drug: MIL62
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: MIL62 — Phase 1b: Participants will receive intravenous (IV) infusions of MIL62 at doses of 500 mg or 1000 mg on Week (W) 1 Day (D) 1, W3D1, W25D1, W27D1, W53D1, W79D1, W105D1, W131D1, W157D1, W183D1, and W209D1. Participants initially assigned to the 500 mg dose group who exhibit good tolerance may be escalated to the 1000 mg dose starting from W25D1.
  Phase 3 (Randomised Controlled Period [RCP]): Participants will receive IV MIL62 1000 mg or placebo matched to MIL62 on W1D1, W3D1, W25D1, and W27D1. The administration protocol for placebo is identical to that of MIL62.
  Phase 3 (Open-Label Period [OLP]): Participants who enter the OLP will receive IV MIL62 1000 mg on W1D1, W27D1, W53D1, W79D1, W105D1, and W131D1, along with matching placebo on W3D1.
  Arms: MIL62
Other: Placebo — Phase 3 (RCP): Participants will receive IV placebo matched to MIL62 on W1D1, W3D1, W25D1, and W27D1.
  Phase 3 (OLP): Participants entering the OLP will receive IV MIL62 1000 mg on W1D1, W3D1, W27D1, W53D1, W79D1, W105D1, and W131D1.
  Arms: Placebo

SUMMARY:
This study will evaluate the safety and efficacy of MIL62 in patients with Neuromyelitis Optica Spectrum Disorder.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who meet the diagnostic criteria for NMOSD established by the International Panel for NMO Diagnosis (IPND) in 2015 and are seropositive for AQP4-IgG.
2. Male or female patients aged 18 to 70 years, inclusive of the endpoints..
3. Expanded Disability Status Scale(EDSS) score ≤ 7.
4. Phase Ib: At least 1 attack of NMOSD requiring rescue treatment within 2 years prior to screening. Phase III: At least 1 attack of NMOSD requiring rescue treatment within 1 year prior to screening; or at least 2 attacks of NMOSD requiring rescue treatment within 2 years prior to screening, including the first attack.
5. Glucocorticoid treatment prior to screening is allowed, and within 14 days before the first administration, the dose should be ≤20 mg/day of prednisone or its equivalent dose of glucocorticoids.
6. Patients who had an attack of the disease before screening must have stable or improved attack symptoms for at least 4 weeks prior to the first administration.
7. Voluntarily sign the informed consent form.

Exclusion Criteria:

1. Subjects who have received Rituximab, Inebilizumab, Ozanimod, Telitacicept, or any B-cell depleting drugs within 6 months prior to the screening period are allowed to enroll if their CD19 or CD20 positive B-cell counts are above the lower limit of normal; or if their CD4 positive T-lymphocyte counts are < 200 cells/μL.
2. Having used Tocilizumab, Satralizumab, Eculizumab, Efgartigimod, or other non-B-cell depleting biological agents with therapeutic effects on NMOSD, or mitoxantrone, or alkylating agents such as cyclophosphamide within 3 months prior to the first administration.
3. Phase Ib: Subjects who have used immunosuppressants such as azathioprine, mycophenolate mofetil, tacrolimus, cyclosporine, methotrexate, and cyclophosphamide before the first administration are eligible for enrollment, provided that the interval since discontinuing the drugs exceeds 5 times their half-life. Phase III: Subjects who have used immunosuppressants other than glucocorticoids within 1 month prior to the first administration, including but not limited to azathioprine, mycophenolate mofetil, tacrolimus, cyclosporine, and methotrexate, are excluded (exclusion is not required if the continuous use duration is ≤7 days).
4. Within 28 days prior to the first administration, plasma exchange (PE), moderate blood transfusion, or immunomodulatory drugs such as interferon β, interferon γ, or intravenous immunoglobulin (IVIG) have been used.
5. Live vaccines or attenuated vaccines were administered within 28 days prior to the first dose.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2022-08-18 (Actual); Primary Completion 2025-02-21 (Actual); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Phase 1b: The incidence and severity of all adverse events (AE) | Up to Week 234
Phase 3: Time to First Adjudicated Relapse (TFR) during RCP. | Up to 52 weeks
  The time from the date of randomization to the date of the first clinical relapse as assessed by the Clinical Endpoint Committee(CEC). The criteria for NMOSD relapse are the occurrence of new objective neurological symptoms or worsening of objective neurological symptoms; meeting any one of the relapse criteria specified in the protocol is sufficient.

SECONDARY OUTCOMES:
Time to first adjudicated relapse | Up to Week 208
Annualized relapse rate | Up to Week 208
Change from baseline of Expanded Disability Status Scale (EDSS) score | Up to Week 208
Annualized cumulative active lesions rate on MRI | Up to Week 208
Annualised NMOSD-related inpatient hospitalisation rate. | Up to Week 208
Mean Change in T-score from Baseline in the EQ5D Scale. | Up to Week 208
Percentage of Participants with Adverse Events (AEs). | Up to Week 208
  Severity Determined According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0
Peripheral B-cell Counts at Specified Timepoints. | Up to Week 208

CONTACTS AND LOCATIONS:
Locations (1):
- Ethics Committee of Chinese PLA General Hosptial, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No